CLINICAL TRIAL: NCT05434884
Title: Clinical Performance of Two CAD/CAM Fabricated Ceramic Restorations With Different Preparation Designs for Rehabilitation Of Permanent First Molars Affected With Molar Incisor Hypomineralisation (MIH): Clinical Randomized Trial
Brief Title: Clinical Performance of Two Cad-cam Fabricated Ceramic Restoration in Teeth Affected With MIH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Collaborators: Altura (Industry)
Responsible Party: Principal Investigator, sara nabil, Lecturer of pediatric dentistry, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AlAzharUniversity
Record Dates: First submitted 2022-02-10; First posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Molar Incisor Hypomineralization
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial (RCT)
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OV group (Experimental): Patients will receive occlusal veneer restorations
  Interventions: Procedure: occlusal veneer restorations
- EN group (Experimental): Patients will receive endocrown restorations
  Interventions: Procedure: endocrown restorations

INTERVENTIONS:
Procedure: occlusal veneer restorations — occlusal veneer preparation with circumferential chamfer finish line and proximal slot " proposed modified occlusal veneer design" for rehabilitation of moderate level of permanent first molars. OrPatients will receive endocrown restorations for rehabilitation of sever level of permanent first molars
  Arms: OV group
Procedure: endocrown restorations — endocrown restorations
  Arms: EN group

SUMMARY:
This study will be performed to evaluate the clinical performance (Plaque accumulation, fracture of (restoration or tooth), postoperative sensitivity, secondary caries, marginal fit and discoloration) of two CAD/CAM fabricated ceramic restorations (zirconia-reinforced lithium silicate glass ceramic and hybrid ceramic) with different preparation designs (modified occlusal veneer and endocrown) for rehabilitation of permanent first molars affected with different severity level of molar incisor hypomineralisation (MIH), evaluated at different time periods

DETAILED DESCRIPTION:
Clinical evaluation of all restorations will be performed according to:

- Modified United States Public Health Service (USPHS) Ryge Criteria, at base line (1 week), 3, 6 and 12 months after cementation.

ELIGIBILITY:
Inclusion Criteria:-

* Patient from 8 to 13 years
* permanent first molar tooth affected with different severity levels of MIH
* Ability to physically and psychologically tolerate conventional restorative procedures.

Exclusion Criteria:.

* Patients have active periodontal diseases.
* Patient with poor oral hygiene and motivation.
* Patient with psychiatric problems or unrealistic expectations

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
retention | 1 year
  Clinical evaluation of all restorations will be performed according to:
  - Modified United States Public Health Service (USPHS) Ryge Criteria,at12 month after cementation
marginal integrity | 6 months
  Clinical evaluation of all restorations will be performed according to:
  - Modified United States Public Health Service (USPHS) Ryge Criteria, at 6 months after cementation
colour stability | 12 months
  Clinical evaluation of all restorations will be performed according to:
  - Modified United States Public Health Service (USPHS) Ryge Criteria, at 12 months after cementation
Elimination of sensitivity | 3 months
  Clinical evaluation of all restorations will be performed according to:
  - Modified United States Public Health Service (USPHS) Ryge Criteria, at 3, months after cementation

CONTACTS AND LOCATIONS:
Overall Officials: Mona Hossam, professor, Study Director — doctor
Locations (1):
- Dr.sara nabil, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
sharing primary results only